CLINICAL TRIAL: NCT05037162
Title: A Phase IIb, Double Blind, Placebo-controlled Clinical Study Designed to Evaluate the Effect of CimetrA in Patients Diagnosed With COVID-19
Brief Title: Study Designed to Evaluate the Effect of CimetrA in Patients Diagnosed With COVID-19
Acronym: CimetrA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MGC Pharmaceuticals d.o.o (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGC-009
Record Dates: First submitted 2021-08-15; First posted 2021-09-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Corona Virus Infection
Keywords: Corona; covid19; COVID-19; coronavirus; corona virus infection; sars-cov-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Blood Coagulation; Vital Signs; Pregnancy Tests; Physical Examination; COVID-19 Testing; Electrocardiography

STUDY DESIGN:
Intervention Model Description: Multi-center multinational-controlled study in Israel, Brazil, Spain, and South-Africa.
  240 adult patients who suffer from moderate COVID-19 infection. Safety will be assessed through collection and analysis of adverse events, blood and urine laboratory assessments and vital signs.
  After Screening visit, the study drug will be administrated twice a day morning and evening (every 12 hours) during (day 1 and day 2) The patients will be randomized in 1:1:1 ratio to study drug (CimetrA) in two dosages in addition to Standard of Care - Arm 1, 2 or (Placebo) in addition to Standard of Care- Arm 3.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study: neither the participants nor the investigators will be aware of arm allocation of each study participant.
  Blindness is important to avoid bias. Monitoring and reporting of the success of blindness are important for the reader's confidence of the trial results. Groups should be marked by capital letter and blindness should maintain throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - CimetrA-1 (Experimental): CimetrA-1, with a total dose containing a combination of Curcumin 40 mg, Boswellia 30 mg and Vitamin C 120 mg in spray administration - divided in 4 separate doses given as an add on therapy, total of 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Diagnostic Test: Biochemistry blood test; Diagnostic Test: Hematology blood test; Diagnostic Test: D-Dimer test (coagulation); Diagnostic Test: Inflammatory markers; Diagnostic Test: Vital signs; Diagnostic Test: VAS scale; Diagnostic Test: WHO Ordinal Score; Diagnostic Test: COVID-19-Related Symptoms assessment; Diagnostic Test: COVID-19-Impact on Quality-of-Life Questionnaire; Diagnostic Test: POST- COVID-19 Functional Status Scale:; Diagnostic Test: Pregnancy test; Diagnostic Test: Physical examination; Diagnostic Test: PK parameters; Diagnostic Test: SARS-CoV-2 test (PCR); Diagnostic Test: ECG; Drug: Treatment administration (twice a day)
- Arm 2 - CimetrA-2 (Experimental): CimetrA-2, with a total dose containing a combination of Curcumin 28 mg, Boswellia 21 mg and Vitamin C 84 mg in spray administration - divided in 4 separate doses given as an add on therapy, total of 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Diagnostic Test: Biochemistry blood test; Diagnostic Test: Hematology blood test; Diagnostic Test: D-Dimer test (coagulation); Diagnostic Test: Inflammatory markers; Diagnostic Test: Vital signs; Diagnostic Test: VAS scale; Diagnostic Test: WHO Ordinal Score; Diagnostic Test: COVID-19-Related Symptoms assessment; Diagnostic Test: COVID-19-Impact on Quality-of-Life Questionnaire; Diagnostic Test: POST- COVID-19 Functional Status Scale:; Diagnostic Test: Pregnancy test; Diagnostic Test: Physical examination; Diagnostic Test: PK parameters; Diagnostic Test: SARS-CoV-2 test (PCR); Diagnostic Test: ECG; Drug: Treatment administration (twice a day)
- Arm 3 - Placebo (Placebo Comparator): Placebo, composed of the same solvent but without active ingredients, given as an add on therapy in spray administration, total of 4 doses over 48 hours (day 1 and day 2), twice a day (morning and evening).
  Interventions: Diagnostic Test: Biochemistry blood test; Diagnostic Test: Hematology blood test; Diagnostic Test: D-Dimer test (coagulation); Diagnostic Test: Inflammatory markers; Diagnostic Test: Vital signs; Diagnostic Test: VAS scale; Diagnostic Test: WHO Ordinal Score; Diagnostic Test: COVID-19-Related Symptoms assessment; Diagnostic Test: COVID-19-Impact on Quality-of-Life Questionnaire; Diagnostic Test: POST- COVID-19 Functional Status Scale:; Diagnostic Test: Pregnancy test; Diagnostic Test: Physical examination; Diagnostic Test: PK parameters; Diagnostic Test: SARS-CoV-2 test (PCR); Diagnostic Test: ECG; Drug: Treatment administration (twice a day)

INTERVENTIONS:
Diagnostic Test: Biochemistry blood test — preformed on days 1-14 and day 28. Sodium (Na), Potassium (K), Chloride (Cl), Creatinine, Glucose, Urea, Albumin, Calcium total, Alkaline Phosphatase (ALP), ALT, AST, Total Bilirubin, Direct Bilirubin, LDH, Total Protein, Uric Acid, CRP, and Lipid Profile (including Total Cholesterol, HDL,
Diagnostic Test: Hematology blood test — preformed on days 1-14 and day 28. complete CBC.
Diagnostic Test: D-Dimer test (coagulation) — performed on days 1,2,7,14 and 28.
Diagnostic Test: Inflammatory markers — performed on days 1-7, 14 and 28. IL-6, IL-1β, IL-12, TNF α, IFN-γ
Diagnostic Test: Vital signs — performed on days 1-14 and day 28. blood pressure, pulse, weight, weight, body temperature (PO), saturation, respiratory rate.
Diagnostic Test: VAS scale — performed on all study visits. score: 0-10 ; a higher score indicates a higher pain level.
Diagnostic Test: WHO Ordinal Score — performed on days 1,7,14 and 28. score: 0-3 ; a higher score indicates more symptoms.
Diagnostic Test: COVID-19-Related Symptoms assessment — performed on days 1,7,14,21 and 28. score: 0-3 ; a higher score indicates more symptoms.
Diagnostic Test: COVID-19-Impact on Quality-of-Life Questionnaire — performed on days 1,7,14,21 and 28. score: 1-5 ; a higher score indicates a lower quality of life.
Diagnostic Test: POST- COVID-19 Functional Status Scale: — performed on day 28. score: 0-3 ; a higher score indicates better recovery.
Diagnostic Test: Pregnancy test — performed on days 1 and 28. women of childbearing potential must undergo a urine pregnancy test.
Diagnostic Test: Physical examination — performed on days 1-14 and day 28. a full examination by a doctor.
Diagnostic Test: PK parameters — performed on day 1. will be performed only on 14 patients that will agree to participate in the PK analysis (only for Brazil,Spain).
  The PK will be performed only for the first dose of drug, after patient received the first dose (5 puffs) the study staff need to follow the table below.
  For each test, approximately 5 ml of blood will be drawn (equivalent to one teaspoon)
Diagnostic Test: SARS-CoV-2 test (PCR) — performed on days 1,14 and 28.
Diagnostic Test: ECG — performed on days 1 and 28.
Drug: Treatment administration (twice a day) — performed on days 1 and 2. twice a day, morning, and evening 1:1:1 ratio to study drug (CimetrA-1) (Arm 1) or study drug (CimetrA-2) or to Placebo (Arm 3)

SUMMARY:
Multi-center multinational-controlled study in Israel, Brazil, Spain, and South-Africa.

240 adult patients who suffer from moderate COVID-19 infection. Safety will be assessed through collection and analysis of adverse events, blood and urine laboratory assessments and vital signs.

After Screening visit, the study drug will be administrated twice a day morning and evening (every 12 hours) during (day 1 and day 2) The patients will be randomized in 1:1:1 ratio to study drug (CimetrA) in two dosages in addition to Standard of Care - Arm 1, 2 or (Placebo) in addition to Standard of Care- Arm 3.

DETAILED DESCRIPTION:
A preparation of CimertA (Botanical Drug), comprising Curcumin, Boswellia, and Vitamin C in a nanoparticular formulation, is proposed as a treatment for the disease associated with the novel corona virus SARS-CoV-2. This initiative is presented under the urgent circumstances of the fulminant pandemic caused by this lethal disease, which is known as COVID-19 and has spread across the globe causing death and disrupting the normal function of modern society. The grounds for the proposal are rooted in existing knowledge on the components and pharmacological features of this formulation and their relevance to the current understanding of the disease process being addressed.

The breakout of a lethal pneumonia in the city of Wuhan, China, towards the end of 2019, has led to the characterization of the new coronavirus related disease COVID-19. Its prominent features include a high rate of person-to-person transmission, a substantial risk of developing a lethal respiratory syndrome and potential failure of additional organs. Risk factors for a life-threatening clinical course have been identified, including advanced age and assorted comorbidities, such as cardiovascular disease, diabetes mellitus, hypertension, cancer. However, individuals devoid of any of the recognized risk factors are not immune to the severe manifestation of the disease and once infected carry a certain risk of mortality which has been calculated in Italy at circa 2%.

CoV is an enveloped, positive-sense single-stranded RNA (ss-RNA) virus belonging to the Coronaviridae family. The severe acute respiratory syndrome associated coronavirus disease 2019 (COVID-19) illness is a syndrome of viral replication in concert with a host inflammatory response. The cytokine storm and viral evasion of cellular immune responses may play an equally important role in the pathogenesis, clinical manifestation, and outcomes of COVID-19. Systemic proinflammatory cytokines and biomarkers are elevated as the disease progresses towards its advanced stages, and correlate with worse chances of survival.

SARS-CoV-2 activates the innate immune system and results in a release of a large number of cytokines, including IL-6, which can increase vascular permeability and cause a migration of fluid and blood cells into the alveoli as well as the consequent symptoms such as dyspnea and respiratory failure. The higher mortality is being linked to the result of ARDS (acute respiratory distress syndrome) aggravation and the tissue damage that can result in organ-failure and/or death.

Serum cytokine levels that are elevated in patients with Covid-19-associated cytokine storm include interleukin-1β, interleukin-6, IP-10, TNF, interferon-γ, macrophage inflammatory protein (MIP) 1α and 1β, and VEGF. Higher interleukin-6 levels are strongly associated with shorter survival. The relative frequencies of circulating activated CD4+ and CD8+ T cells and plasma blasts are increased in Covid-19. In addition to the elevated systemic cytokine levels and activated immune cells, several clinical and laboratory abnormalities, such as elevated CRP and d-dimer levels, hypoalbuminemia, renal dysfunction, and effusions, are also observed in Covid-19, as they are in cytokine storm disorders. Laboratory test results reflecting hyperinflammation and tissue damage were found to predict worsening outcomes in Covid-19.

CimetrA, comprising Curcumin, Boswellia, and Vitamin C in a nanoparticular formulation, was studied on patients with the novel corona virus SARS-CoV-2 in randomized double blind control Phase II study (MGC-006 - under a previous product name - ArtemiC). The study product demonstrated excellent safety and efficacy profiles.

In the in vitro clinical trial CimetrA demonstrated the ability to reduce cytokines elevation in PBMC induced cell tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by PCR test SARS-CoV-2 infection (according to nationally authorized laboratory criteria)
2. Hospitalized patient with COVID-19 of moderate stable or worsening severity not requiring ICU admission (defined by NIH criteria - fever, cough, dyspnea, fast breathing, but no signs of severe pneumonia, including SpO2 ≥ 94% on room air).
3. Age: 18 years old and above.
4. Subjects must be hospitalized
5. Ability to receive treatment by spray into the oral cavity

Exclusion Criteria:

1. Tube feeding or parenteral nutrition.
2. Patients with scores 5 or above per the Ordinal Scale for Clinical Improvement published by the WHO. (i.e., who need oxygen supply beyond use of nozzles or simple mask)
3. Need for admission to ICU during the present hospitalization at any time prior to completion of the recruitment to the study.
4. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in WHO Ordinal Scale for clinical improvement | up to 28 days
  measured on days 1, 7, 14, 28 numerical value to assess the health status of the participant , scale is between 0-8 , The higher score means the worse outcome .
Change in COVID-19-Related Symptoms score | up to 28 days
  measured on days 1,7, 14, 28 numerical value to assess the COVID-19-Related symptoms of participant scale is between 0-3, The higher score means the worse outcome .
  score 0-3; higher score indicates worse outcome.
Safety endpoint: will be assessed through collection and analysis of adverse events | up to 28 days
  Data management team will assess and review the AE's and SAE'S.
Safety endpoint: will be assessed through collection and analysis of blood laboratory test. | up to 28 days
  Data management team will assess and review the lab test results (blood), assessment will be compared to the normal range. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint: will be assessed through collection and analysis of urine laboratory test. | up to 28 days
  Data management team will assess and review the lab test results (urine), assessment will be compared to the normal range. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint: will be assessed through collection and analysis of blood preasure | up to 28 days
  units: BPM (beats per minute) Data management team will assess and review the vital signs : blood pressure [mm Hg], saturation [%], body temperature [C] , Each category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint: will be assessed through collection and analysis of blood satturation | up to 28 days
  units: %O2 Data management team will assess and review the vital signs : blood pressure [mm Hg], saturation [%], body temperature [C] , Each category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint: will be assessed through collection and analysis of body temperature | up to 28 days
  units: celsius degrees Data management team will assess and review the vital signs : blood pressure [mm Hg], saturation [%], body temperature [C] , Each category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition

SECONDARY OUTCOMES:
Number of participants with depending on oxygen supplementation through day 28 since onset of symptoms | up to 28 days
Change in inflammatory marker levels - IL-6, IL-1β, IL-12, TNF α, IFN-γ, CRP, NLR (Neutrophil / Lymphocyte ratio) at days 1, 2, 4, 7, compared to baseline | up to 7 days
Pharmacokinetic profile of the study drug | on day 1 through 24 Hrs
  Measurements :
  CMAX elimination rate constant (denoted as K) half-life (t 1/2) apparent volume of distribution (V d) total clearance rate (CL). AUC
Pharmacokinetic profile of the study drug - maximal concentartion | on day 1 through 24 Hrs
  CMAX measurement (mg/ml)
Pharmacokinetic profile of the study drug - elimination rate constant (denoted as K) | on day 1 through 24 Hrs
  (mg/ml/min)
Pharmacokinetic profile of the study drug - half-life | on day 1 through 24 Hrs
  half-life t 1/2 (Min)
Pharmacokinetic profile of the study drug - apparent volume of distribution | on day 1 through 24 Hrs
  apparent volume of distribution V d (mL)
Pharmacokinetic profile of the study drug - total clearance rate | on day 1 through 24 Hrs
  total clearance rate CL (min/mg)
Pharmacokinetic profile of the study drug - AUC | on day 1 through 24 Hrs
  AUC (min)
duration of mechanical ventilation | up to 28 days
  in days
Incidence of Intensive Care Unit (ICU) stay during COVID-19 complication | up to 28 days
Percentage of participants with definite or probable drug related adverse events | up to 28 days
Long term adverse events of COVID-19 on Day 28 | up to 28 days
  The Outcome will Measure the number of patients who recovered from covid_19 , but still have adverse events.
The Impact covid_19 on Quality of life of patients on Days 1, 14 and 28. | up to 28 days
  numerical value to assess the the impact of covid_19 on the quality life of the participant, scale is between 1-5, as expressed in the subject's subjective perception, The higher score is more important.
Course of change in D Dimer levels compared to baseline | up to 28 days
Occurrence of secondary infections | up to 28 days
Incidence of mechanical ventilation | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nadaf, Study Director — Galilee CBR - CRO
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No